CLINICAL TRIAL: NCT03398733
Title: Preoperative CPAP Treatment on Perioperative Outcomes in Rheumatic Valvular Heart Disease Patients With OSA
Brief Title: CPAP Treatment and Postoperative Outcomes in Patients With Rheumatic Valvular Heart Disease
Acronym: CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ning Ding, Principal Investigator, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-SR-040
Record Dates: First submitted 2018-01-01; First posted 2018-01-12 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Rheumatic Valvular Heart Disease; Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; heart valve replacement; CPAP treatment
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: A total of 200 patients with rheumatic valvular heart disease waiting for heart valve replacement were screened for obstructive sleep apnea (OSA). Of them, 30 OSA patients were enrolled and randomly received CPAP treatment and non-CPAP treatment (15:15 patients).The CPAP treatment group received both baseline and CPAP treatment for 7 days preoperatively. The non-CPAP treatment group only received baseline treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- continuous positive airway pressure (Other): The CPAP treatment group received both baseline and CPAP treatment for 7 days preoperatively.
  Interventions: Device: continuous positive airway pressure

INTERVENTIONS:
Device: continuous positive airway pressure — The CPAP treatment group received both baseline and CPAP treatment for 7 days preoperatively. The non-CPAP treatment group only received baseline treatment.

SUMMARY:
The prevalence of OSA (Obstructive sleep apnea，OSA) is 2%-4% in general population and 16%-47% in surgical-heart failure patients. Our previous study found that OSA was associated with the increasing incidence of perioperative adverse events.The continuous positive airway pressure (CPAP), as the standard treatment for OSA, is extensively applied clinically. The previous study reported that postoperative AHI was reduced and SPO2 was increased by CPAP treatment. However, whether CPAP treatment can improve OSA postoperative and related adverse events or not in patients with rheumatic valvular heart diseases (RVHD) were not reported.The purpose of this study is to observe the effective of preoperative CPAP on postoperative sleep parameters and adverse events, such as AHI changes, duration of ICU stay and duration of mechanical ventilation.

DETAILED DESCRIPTION:
Between December 1, 2017 and June 30 2019, 200 patients with chronic heart failure caused by rheumatic valvular heart disease waiting for heart valve replacement in Department of Cardiovascular Surgery were screened for obstructive sleep apnea (OSA) by full-night polysomnography (PSG). Of them, 30 OSA patients were enrolled and randomly received CPAP treatment and non-CPAP treatment (15:15).

The CPAP treatment group received both baseline and CPAP treatment. The full-night CPAP treatment was conducted from 21:00 pm to 6:00 am for 7 days preoperatively. The non-CPAP treatment group received baseline treatment.

Preoperative Sleep parameters (AHI, mean and lowest SPO2) and clinical evaluations including NYHA class, electrocardiographic, echocardiographic, arterial blood gas analysis findings, baseline medication, and 6-minute walk test were recorded.

Operation related parameters such as duration of operation, duration of cardiopulmonary bypass and bleeding volume were recorded.

Postoperative adverse events such as duration of ICU stay, postoperative duration of mechanical ventilation, pacemaker use, complicated infection and reintubation are recorded.

A PSG was re-examined before discharge from hospital. The changes of AHI, mean and lowest SPO2 between pre- and post-operative PSG parameters were calculated.

The operation related parameters, postoperative adverse events and the changes of sleep parameters were compared between CPAP and non-CPAP patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-75 years.
2. Patients with rheumatic valvular heart disease.
3. Patients combined with obstructive sleep apnea (apnea-hypopnea index >=5/h).
4. Received heart valve replacement surgery.
5. The enrolled patients having received patients' informed consent.

Exclusion Criteria:

1. History of stroke or clinical signs of peripheral or central nervous system disorders.
2. History of Chronic obstructive pulmonary disease or asthma.
3. Enrolment in another clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
apnea-hypopnea index (AHI) | 2 weeks,depends on length of hospital stay
  The changes of apnea-hypopnea index pre- and post-operative were compared between CPAP and non-CPAP patients.
duration of ICU stay | 3 days, depends on the patient's recovery
  Postoperative duration of ICU stay was compared between CPAP and non-CPAP patients.
length of mechanical ventilation | 1 day, depends on the patient's recovery
  Postoperative length of mechanical ventilation was compared between CPAP and non-CPAP patients.

SECONDARY OUTCOMES:
mean and lowest SPO2 | 2 weeks,depends on length of hospital stay
  The changes of mean and lowest SPO2 pre- and post-operative were compared between CPAP and non-CPAP patients
pacemaker use | 3 days, depends on the patient's recovery
  Postoperative pacemaker use was compared between CPAP and non-CPAP patients.
complicated infection and reintubation | 3 days, depends on the patient's recovery
  Postoperative complicated infection and reintubation were compared between CPAP and non-CPAP patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Ding, MD, PhD, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared. The informed consent will be ansigned before enrolled in the study and ensured to keep personal information confidential.

REFERENCES:
- [Background] Ding N, Ni BQ, Wang H, Ding WX, Xue R, Lin W, Kai Z, Zhang SJ, Zhang XL. Obstructive Sleep Apnea Increases the Perioperative Risk of Cardiac Valve Replacement Surgery: A Prospective Single-Center Study. J Clin Sleep Med. 2016 Oct 15;12(10):1331-1337. doi: 10.5664/jcsm.6182. PMID 27448416
- [Derived] Su M, Lin W, Xu Q, Ni B, Zhang X, Zhang S, Ding N. Impact of 1-week preoperative auto-CPAP treatment on postoperative outcomes in patients undergoing heart valve replacement surgery: a prospective randomized controlled trial. Front Neurol. 2023 Jun 5;14:1152168. doi: 10.3389/fneur.2023.1152168. eCollection 2023. PMID 37342775